CLINICAL TRIAL: NCT02177552
Title: Study Assessing the Effects of Chemotherapy in Advanced Esophagogastric Adenocarcinoma - Carboplatin, Docetaxel and Capecitabine (CTX) or Epirubicin, Oxaliplatin and Capecitabine: a Randomised Phase 2 Trial.
Brief Title: Study Assessing the Effects of Chemotherapy in Advanced Esophagogastric Adenocarcinoma
Acronym: SEED
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Peter Clausager Petersen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01052014; 2014-000127-24 (EudraCT Number)
Record Dates: First submitted 2014-06-18; First posted 2014-06-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Neoplasms; Stomach Neoplasms
Keywords: Esophageal cancer; Gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Carboplatin; Docetaxel; Capecitabine; Epirubicin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental chemotherapy (Experimental): Intravenous carboplatin (C) AUC5 day 1 plus intravenous docetaxel (T) 60 mg/m2 day 1 plus oral capecitabine (X) 1000 mg/m2 twice daily from day 1-14, every 4 weeks.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Drug: Capecitabine
- Standard chemotherapy (Other): Intravenous epirubicin (E) 50 mg/m2 day 1 plus intravenous oxaliplatin (O) 130 mg/m2 day 1 plus oral capecitabine (X) 625 mg/m2 twice daily continuously, every 3 weeks
  Interventions: Drug: Capecitabine; Drug: Epirubicin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Carboplatin
  Arms: Experimental chemotherapy
Drug: Docetaxel
  Arms: Experimental chemotherapy
Drug: Capecitabine
Drug: Epirubicin
  Arms: Standard chemotherapy
Drug: Oxaliplatin
  Arms: Standard chemotherapy

SUMMARY:
The main purpose of this study is to determine the effects of treatment with carboplatin, docetaxel and capecitabine in patients with incurable cancer of the esophagus or stomach.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with histologically verified, unresectable or metastatic, HER2-negative, adenocarcinoma of the esophagus or stomach
* Men or women less than 80 years of age
* Performance status 0 or 1
* Life expectancy >12 weeks
* Adequate organ-function
* Written informed consent

Key Exclusion Criteria:

* Prior chemotherapy for adenocarcinoma of the esophagus or stomach if the chemotherapy-free interval is less than 6 months
* Progression on first-line chemotherapy for unresectable or metastatic adenocarcinoma of the esophagus or stomach
* Chemotherapy with epirubicin, oxaliplatin, carboplatin, cisplatin or docetaxel less than 6 months before study entry
* Prior cumulative dose of >300 mg/m2 of epirubicin
* Grade ≥ 2 side-effects from previous chemotherapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants alive one year after randomisation | Three and a half years

SECONDARY OUTCOMES:
Time to progression or death due to any cause | Three and a half years
Number of participants with grade 3 and 4 toxicities caused by treatments | Day 1 of every cycle and 30 days after completion of treatment
Time until death due to any cause | Three and a half years
Changes in quality-of-life | Three and a half years
The proportion of participants who have carboplatin, docetaxel and capecitabine re-induced | Five years
Registration of further lines of therapy | Five years

OTHER OUTCOMES:
Analysis of cmet by immunohistochemistry | Three and a half years
  Analysis of archived tumour tissue (primary biopsy, previous surgical resection specimen if available) and metastatic tumour tissue for consenting subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Petersen, MD, Principal Investigator — Finsen Center, Rigshospitalet
Locations (1):
- Finsen Center, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Petersen PC, Petersen LN, Vogelius I, Bjerregaard JK, Baeksgaard L. A randomized phase 2 trial of first-line docetaxel, carboplatin, capecitabine (CTX) and epirubicin, oxaliplatin, capecitabine (EOX) in advanced esophagogastric adenocarcinoma. Acta Oncol. 2021 Jul;60(7):948-953. doi: 10.1080/0284186X.2021.1928281. Epub 2021 Jun 4. PMID 34086514